CLINICAL TRIAL: NCT00474396
Title: Dietary Interventions Evaluating Transport of Uric Acid Across the Tubules
Acronym: dietUAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 04-1094
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2007-05-16 (Estimated); Status verified 2007-05

CONDITIONS: Healthy
Keywords: Uric acid; Dairy; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Low fat dairy diet

SUMMARY:
The purpose of the study is to determine whether low fat dairy diet reduces serum uric acid levels.

DETAILED DESCRIPTION:
Uric acid plays a role not only in the pathogenesis of gout but is also a predictor of cardiovascular disease, hypertension and renal disease in man. We have identified the human urate ion channel transporter (hUAT), located in the proximal convoluted tubule of the kidney that is involved in both the secretion and reabsorption of urate across the tubule. This channel has a unique lectin binding site that in in-vitro studies, has been found to be modulated by glucose, galactose and lactose. We have also identified a mutation (G/A polymorphism) in our laboratory, that in in-vitro studies has demonstrated diminished hUAT channel activity. Cross-sectional studies have earlier shown that uric acid levels vary with serum glucose levels. Studies have also reported that a low-fat dairy diet reduces the incidence of gout, while others have shown that this diet reduces blood pressure significantly when compared with a non-dairy diet. We hypothesize that the effect of blood glucose levels in lowering uric acid levels is through the regulation of hUAT channel activity. We also hypothesize that a low-fat dairy diet reduces serum uric acid levels through hUAT regulation leading to a decrease in the incidence of gout and a reduction in blood pressure levels. In our proposed randomized, controlled, cross-over trial in healthy adult volunteers, we aim to study the effect of a low-fat dairy diet and a non-dairy diet on serum uric acid levels, the renal fractional excretion of uric acid and blood pressure. We will also study the effect of an acute intravenous infusion of glucose on these parameters. DNA analysis for hUAT mutations of study subjects will be done to assess if there is a blunted response of hUAT activity in subjects with the polymorphism as compared to normal individuals.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy adult volunteers

  * Coronary artery disease
  * Glucose intolerance or Diabetes(a fasting blood sugar of less than 100 mg/dl as per the American Diabetes Association guidelines)
  * CHF
  * Gout
  * Lactose intolerance
  * Milk allergy
  * Women who are pregnant or lactating
  * Subjects who are on any medications except birth control pills
  * Subjects who drink more than 3 servings of beer or liquor per week.
  * Normal blood pressure ( less than 120 mmHg systolic and 80 mmHg diastolic)
  * Normal serum UA levels
  * Normal renal funcion (calculated GFR >90ml/min)

Exclusion Criteria:

* • Coronary artery disease

  * Glucose intolerance or Diabetes(a fasting blood sugar of less than 100 mg/dl as per the American Diabetes Association guidelines)
  * CHF
  * Gout
  * Lactose intolerance
  * Milk allergy
  * Women who are pregnant or lactating
  * Subjects who are on any medications except birth control pills
  * Subjects who drink more than 3 servings of beer or liquor per week

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2005-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Lowering of serum uric acid levels

SECONDARY OUTCOMES:
Lowering of the fractional excretion of uric acid and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Rafey, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Background] Rafey MA, Lipkowitz MS, Leal-Pinto E, Abramson RG. Uric acid transport. Curr Opin Nephrol Hypertens. 2003 Sep;12(5):511-6. doi: 10.1097/00041552-200309000-00005. PMID 12920398
- [Background] Choi HK, Atkinson K, Karlson EW, Willett W, Curhan G. Purine-rich foods, dairy and protein intake, and the risk of gout in men. N Engl J Med. 2004 Mar 11;350(11):1093-103. doi: 10.1056/NEJMoa035700. PMID 15014182
- [Background] Appel LJ, Moore TJ, Obarzanek E, Vollmer WM, Svetkey LP, Sacks FM, Bray GA, Vogt TM, Cutler JA, Windhauser MM, Lin PH, Karanja N. A clinical trial of the effects of dietary patterns on blood pressure. DASH Collaborative Research Group. N Engl J Med. 1997 Apr 17;336(16):1117-24. doi: 10.1056/NEJM199704173361601. PMID 9099655